CLINICAL TRIAL: NCT04105075
Title: Features of Chronic Obstructive Pulmonary Disease Clinical Course in Obese Patients
Brief Title: COPD in Obese Patients
Status: Completed | Type: Observational
Sponsor: Voronezh N.N. Burdenko State Medical Academy (Other)
Responsible Party: Sponsor
Other Study IDs: YSShkatova
Record Dates: First submitted 2019-09-22; First posted 2019-09-26 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Copd; Obese; Obesity, Abdominal
Keywords: spirometry; inflammation; copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity; Obesity, Abdominal; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COPD and obesity: Patients consented to have a blood sample taken
- Normal body weight patients with COPD: Patients consented to have a blood sample taken

SUMMARY:
The study included 176 patients with COPD. The first group included 88 normal weight patients with COPD: 71 men and 17 women, mean age 62.40 ± 8.83 years. The second group included 88 patients with COPD and obesity: 64 men and 24 women, mean age 62.94 ± 5.96 years. We assessed the frequency of COPD exacerbations in last 12 months, the severity of symptoms such as dyspnea, sputum production, fatigue. Spirometry, six-minute walk test and analysis of body tissue type composition were performed. BODE index was calculated. Levels of leptin, adiponectin, interleukins-4,6,8,10, interferon-γ, c-reactive protein (CRP), tumor necrosis factor receptor 1 (TNF-R1), tumor necrosis factor receptor 2 (TNF-R2), tumor necrosis factor alpha (TNF-α) were measured in blood serum.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis, informed consent for voluntary participation in the study

Exclusion Criteria:

* patient participation in any interventional study,
* COPD exacerbation,
* concomitant lung diseases, such as confirmed or suspected malignant lung disease or other respiratory disease, such as interstitial pulmonary fibrosis, tuberculosis, sarcoidosis, bronchial asthma, bronchiectasis,
* concomitant diseases of other organs and systems, such as acute cardiovascular diseases, chronic kidney diseases and liver failure.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included 176 patients with COPD. According to the Global Initiative for Chronic Obstructive Lung Disease (GOLD, 2019) classification, all patients belonged to the group D, GOLD 2-4 (GOLD 1 = forced expiratory volume in 1 second (FEV1) ≥ 80% predicted, GOLD 2 = 50 ≤ FEV1 ≤ 80% predicted, GOLD 3 = 30 ≤ FEV1 ≤ 50% predicted, GOLD 4 = FEV1 < 30% predicted). Patients were divided in two groups depending on the body mass index (BMI): 18.5-24.99 kg / m2 - normal weight, 30 kg / m2 and more - obesity. The first group (group 1) included 88 patients with COPD and normal weight: 71 (80.68%) men and 17 (19.32%) women aged from 43 to 72 years (mean age 62.40 ± 8.83 years). The second group (group 2) - 88 patients with COPD and obesity: 64 (72.73%) men and 24 (27.27%) women aged from 50 to 72 years (mean age 62.94 ± 5.96 years).
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Simptoms | 1 year
  dyspnea, sputum production and fatigue
Labotary tests | 1 year
  Levels of interleukins-4,6,8,10, interferon-γ, tumor necrosis factor receptor 1 (TNF-R1), tumor necrosis factor receptor 2 (TNF-R2), tumor necrosis factor alpha (TNF-α) were measured in blood serum (pg / ml)
Spirometry | 1 year
  FEV1, % pred,FVC, % pred.,FEV1/FVC, %
Labotary tests | 1 year
  Levels of leptin (ng / ml) measured in blood serum
Labotary tests | 1 year
  Levels of adiponectin (µg / ml) measured in blood serum

SECONDARY OUTCOMES:
Symptroms and laboratory correlations | 1 year
  Statistical methods allowing to figure out associations and correlations between blood tests and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Budnevsky, Study Director — Voronezh State Medical Univercity
Locations (1):
- Voronezh State Medical University, Voronezh, Russia

IPD SHARING:
Plan to Share IPD: No